CLINICAL TRIAL: NCT00819429
Title: A Nutritional and Social Skills Intervention on Conduct Disorder and Hyperactivity
Brief Title: Supplements and Social Skills Intervention Study
Acronym: SASSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Healthcare Group, Singapore (Other Government)
Collaborators: University of Pennsylvania (Other); National University of Singapore (Other); Duke-NUS Graduate Medical School (Other); Alexandra Hospital (Other); Singapore Institute for Clinical Studies (Other); Nanyang Technological University (Other)
Responsible Party: Principal Investigator, A/Prof Daniel Fung Shuen Sheng, Chairman Medical Board, National Healthcare Group, Singapore
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMRC/1170/2008; DSRB: A/08/410 (Other: NHG Singapore); CRC: 240/2008 (Other: Institute of Mental Health); CTC: 0800590 (Other: Health Sciences Authority)
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Conduct Disorder; Attention Deficit Hyperactivity Disorder; Oppositional Defiant Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Conduct Disorder; Oppositional Defiant Disorder; Omega 3 Supplements; Social Skills Training; Dietary Intake; Aggression; Nutrition; Disruptive Behaviors Disorder
MeSH Terms: conditions — Conduct Disorder; Attention Deficit Disorder with Hyperactivity; Oppositional Defiant Disorder; Aggression | interventions — Docosahexaenoic Acids; Child Guidance Clinics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Omega-3 + Standard treatment
  Children in this group will be given 400 mg of DHA and 600 mg of EPA. Caregivers will be instructed to give two 500mg Omega-3 capsules twice a day, at breakfast and at the evening meal for 6 months. Parents will be seen by the attending on a monthly basis for standard treatment procedure.
  Interventions: Dietary Supplement: Omega-3; Other: Standard Treatment (or TAU in Child Guidance Clinic)
- 2 (Experimental): Social skills + Omega-3 placebo + Standard treatment
  Children in this group will be given two placebo capsules twice daily; at breakfast and at the evening meal for a total period of 6 months. They will also undergo a manualised group social problem solving skills training protocol of 12 weekly 1-hour sessions (Ang & Ooi, 2003a, 2003b). There will be booster sessions scheduled at 3-week intervals after the initial treatment period of 12 weeks, for a total of 4 booster sessions.
  Interventions: Behavioral: Social Skills Training; Other: Standard Treatment (or TAU in Child Guidance Clinic)
- 3 (Experimental): Omega-3 + Social skills + Standard treatment
  Children in this group will receive omega-3 supplement and social skills training on top of standard treatment. Procedures for administration of Omega-3 supplement are similar to those stated in (1) and (2).
  Interventions: Dietary Supplement: Omega-3; Behavioral: Social Skills Training; Other: Standard Treatment (or TAU in Child Guidance Clinic)
- 4 (Placebo Comparator): Omega-3 placebo + Standard treatment.
  Children in this group will receive placebo as well as a course of the standard treatment. Procedure for administering the placebo capsules is similar to that outlined in (2).
  Interventions: Other: Standard Treatment (or TAU in Child Guidance Clinic)

INTERVENTIONS:
Dietary Supplement: Omega-3 — 1000mg of Omega-3 supplement will be given twice a day for a duration of 6 months. All supplements (including placebo) will be administered as two 500mg softgels twice daily, to be taken during breakfast and during the evening meal.
  Arms: 1; 3
Behavioral: Social Skills Training — 1 hourly sessions over 12 weeks duration and 4 booster sessions at 3 weeks intervals. During these 16 sessions, children are taught empathy, pro-social skills, and a variety of positive coping techniques for problem-solving, emotional regulation, conflict resolution, and anger management via the use of practical strategies, materials, activities, role-play and games.
  Arms: 2; 3
Other: Standard Treatment (or TAU in Child Guidance Clinic) — Standard treatment is administered on a monthly basis to the parents of the child participants by the clinicians. Parents will be provided Parent Management Training where they will be taught behaviour and parenting techniques and may be referred to a parent support group. There is clinical pathway for the management of ADHD in our department which will be adhered to (i.e., Clinical Pathway for ADHD).

SUMMARY:
This is a 36-week, randomised, double-blind, placebo-controlled trial. The overarching aim of this study is to assess whether a nutritional intervention (Omega-3 supplement), when combined with a more traditional treatment approach to conduct disorder and Attention Deficit Hyperactivity Disorder (ADHD), is more effective than either approach alone in treating these conditions in children and adolescents. The research questions cannot be answered through alternative means because disruptive behaviour disorders are primarily childhood disorders.

DETAILED DESCRIPTION:
Serious adult crime and violence is a social problem despite decades of intervention and prevention work. One of the reasons for the world-wide failure to prevent this problem stems from (a) a failure to tackle the biological component of the crime/ violence equation in treatment programs, and (b) the failure to tackle this adult condition in its formative childhood origins. Investing modest resources in early biosocial prevention programs could yield enormous long-term financial dividends in terms of the saved legal, medical, social, and psychological costs resulting from adult crime. This initial study would be the first to test the efficacy of conjoint Omega-3 plus social skills training, and the first to identify possible mechanisms by which Omega-3 reduces antisocial behaviour.

A) Initial evidence for effects of Omega-3 supplementation on conduct disorder and Attention Deficit Hyperactivity Disorder (ADHD) B) Moderators of the hypothesised relationship between omega-3 supplementation and conduct disorder C) Social skills training as a treatment for conduct disorder D) The combined effectiveness of omega-3 and social skills training E) Mechanisms of action underlying any treatment effect

The total daily dosages will be 400 mg of DHA and 600 mg of EPA, typical of prior intervention studies of children in the age-range in the proposed study (e.g. Itomura et al. 2005; Richardson & Puri, 2002).

The study involves children and adolescents diagnosed with disruptive behaviour disorder (DBD, i.e. conduct disorder or oppositional defiant disorder) or attention deficit / hyperactivity disorder (ADHD, i.e. combined type or ADHD predominantly inattentive type or ADHD predominantly hyperactive-impulsive type). The overarching aim of this study is to assess whether a nutritional intervention (Omega-3 supplement), when combined with a more traditional treatment approach to conduct disorder and ADHD, is more effective than either approach alone in treating these conditions in children and adolescents. The research questions cannot be answered through alternative means because disruptive behaviour disorders are primarily childhood disorders.

Violence is a world-wide public health problem that has largely defied successful intervention and prevention. The overarching aim of this study is to assess whether a nutritional intervention, when combined with social skills training, is more effective than either approach alone in reducing childhood conduct disorder, the precursor to adult crime and violence. The specific aims are:

Subjects will consist of 600 male and female children seeking treatment at the Child Guidance Clinic.

Subjects given a primary diagnosis by the attending physician of either a disruptive behaviour disorder (DBD, i.e. conduct disorder or oppositional defiant disorder) or attention deficit / hyperactivity disorder (ADHD, i.e. combined type or ADHD predominantly inattentive type or ADHD predominantly hyperactive-impulsive type) will be included.

This a randomised, double-blind, placebo-controlled trial with 4 x 3 x 4 x 2 (4 treatments groups x 3 diagnostic groups x 4 time measurements of an outcome variable x 2 genders) between-subject design to evaluate whether Omega-3 supplement, when combined with social skills training, is more effective than either approach alone in reducing childhood conduct disorder and attention deficit hyperactivity disorder.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between ages 7 and 16 years
* Subjects who fulfils all criteria for a DSM-IV diagnosis of ADHD, conduct disorder, or oppositional defiant disorder
* Subjects with willingness to participate in a randomized, double-blind controlled trial,
* Subjects with complete with written, informed parental consent and assent
* Subjects with IQ of 70 or more

Exclusion Criteria:

* Subjects who have IQ in the below 70
* Subjects who are younger than 7 years old
* Those without written parental consent will not be allowed to participate in the study
* Those with brain pathology such as serious head injury, epilepsy will be excluded

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 282 (Actual)
Dates: Start 2009-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Reactive - Proactive Aggression Questionnaire (RPQ) | 48 weeks
  Changes from baseline to Weeks 12, 24, 36 and 48 in Reactive-Proactive Aggression Questionnaire (Raine et al., 2006) total score

SECONDARY OUTCOMES:
Computerised Diagnostic Interview Schedule for Children - Version IV (C-DISC) | 48 weeks
Clinical Global Assessment Scale | 48 weeks
  Assessment of the participants's level of general functioning using the Children's Global Assessment Scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniel SS Fung, A/Prof, Principal Investigator — Institute of Mental Health, Singapore
Locations (1):
- Child Guidance Clinic, Health Promotion Board, Institute of Mental Health, Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Raine A, Ang RP, Choy O, Hibbeln JR, Ho RM, Lim CG, Lim-Ashworth NSJ, Ling S, Liu JCJ, Ooi YP, Tan YR, Fung DSS. Omega-3 (omega-3) and social skills interventions for reactive aggression and childhood externalizing behavior problems: a randomized, stratified, double-blind, placebo-controlled, factorial trial. Psychol Med. 2019 Jan;49(2):335-344. doi: 10.1017/S0033291718000983. Epub 2018 May 10. PMID 29743128
- [Derived] Liu JC, Raine A, Ang RP, Fung DS. An analysis of blinding success in a randomised controlled trial of fish oil omega-3 fatty acids. Ann Acad Med Singap. 2015 Mar;44(3):85-91. PMID 25882235